CLINICAL TRIAL: NCT05815940
Title: A MOBILE APPLICATION DEVELOPED FOR CHILDREN WITH URINARY INCONTINENCE: PILOT STUDY
Brief Title: A MOBILE APPLICATION DEVELOPED FOR CHILDREN WITH URINARY INCONTINENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Merve Çakırlı, Research Assisstant, Eskisehir Osmangazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EskisehirOU-cakirli-2
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Urinary Incontinence
Keywords: Mobile Application; Child; Quality of Life
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pilot study (Experimental): This was followed by the second phase, during which the mobile application developed was pilot tested with 10 children. Based on the feedback received from the users, the mobile application was finalized.
  Interventions: Behavioral: Mobile Application

INTERVENTIONS:
Behavioral: Mobile Application — a mobile application was developed that can be used by children with urinary incontinence and their parents.

SUMMARY:
The study included 2 stages: In the first, a mobile application with content including urotherapy training and patient follow-up was developed. In the second, a pilot study with the developed mobile application was carried out with 10 children.

DETAILED DESCRIPTION:
The study include two stages. In the first, a mobile application was developed that can be used by children with urinary incontinence and their parents. The mobile application includes the training on urinary incontinence and urotherapy in children as well as all the test results of the child and ensures the follow-up of the children's compliance with the treatment. The developed mobile application is operatable on smartphones and tablets with Android and IOS operating systems.

This was followed by the second phase, during which the mobile application developed was pilot tested with 10 children. Based on the feedback received from the users, the mobile application was finalized.

Mobile application development process

1. Content Creation For Goals
2. Interface design development on MS Word and Photoshop
3. Evaluation by specialists for content and design
4. Converting to mobile application on Android and IOS platforms
5. A pilot study with 10 children to evaluate the usability and suitability of the application
6. Get feedback on the mobile app
7. Based on this feedback, the mobile application was revised.
8. Its final version was created

ELIGIBILITY:
Inclusion Criteria:

* The child has day and/or night urinary incontinence,
* The child is between 7-12 years of age,
* Family members and children can use mobile applications,
* Family members have a smartphone,
* The child and family members volunteers to participate in the study.

Exclusion Criteria:

* The child has a mental or neurological disability,
* The child has a developmental delay,
* The child has previously received treatment for urinary incontinence,
* The child has a communication problem,
* The child has a history of surgery related to the urinary tract,
* The child has a psychiatric diagnosis,
* The child has a urinary tract infection,
* The child has a radiological pathology on ultrasound,
* The child has a diagnosis of neurogenic bladder.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
mobile application development | six months
  a mobile application was developed that can be used by children with urinary incontinence and their parents. The mobile application includes the training on urinary incontinence and urotherapy in children as well as all the test results of the child and ensures the follow-up of the children's compliance with the treatment. The developed mobile application is operatable on smartphones and tablets with Android and IOS operating systems.

SECONDARY OUTCOMES:
pilot tested | one month
  This was followed by the second phase, during which the mobile application developed was pilot tested with 10 children. Based on the feedback received from the users, the mobile application was finalized.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Acikgoz A, Cakirli M, Tokar B, Celik O. SunCloud: A mobile application for children with urinary incontinence. J Eval Clin Pract. 2025 Feb;31(1):e14122. doi: 10.1111/jep.14122. Epub 2024 Aug 7. PMID 39113266